CLINICAL TRIAL: NCT02661399
Title: Investigation of Peripheral Blood Biomarkers Associated With CIPN
Brief Title: Peripheral Blood Biomarkers Associated With CIPN
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Raymond C. Tait, PhD, Professor, St. Louis University
Other Study IDs: 24834
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Peripheral Neuropathy, Secondary to Drugs or Chemicals
Keywords: CIPN
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are doing a research study that will teach us about the tingly pain that people develop when they get chemotherapy.

DETAILED DESCRIPTION:
The investigators are asking for a blood sample, information about patients symptoms during chemotherapy, and past medical history from people who have taken or will take certain types of chemotherapy. The investigators hope to examine blood for proteins that could help us learn which patients get neurological symptoms while getting chemotherapy. The investigators' main research goal is to improve the treatment of patients getting chemotherapy to help their quality of life and/or help to increase the chance of their cancer being cured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a tumor for which Platinums, Vinca Alkaloids, Bortezomib or Taxanes are indicated
* No prior history of diabetic, anatomical or regional neuropathies (except pre-existing CIPN)
* Age ≥ 18 years
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.

Exclusion Criteria:

* Inability to give consent
* Inability to tolerate venipuncture for any reason
* Age < 18 years
* Any known medical, surgical or psychiatric condition that may interfere with the conduct of the study or be detrimental to the donor in the opinion of the PI or caring physician
* Consent Refusal by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have diagnoses which might be treated with CIPN causing therapy, and/or who have CIPN symptoms without potential confounding neuropathies (antecedent diabetic or anatomical peripheral neuropathies).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2017-05-08 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Collection of blood samples, medical history, CIPN symptomology (via questionnaire) and clinical laboratory data for a correlative evaluation of potential CIPN related molecular and cellular variance (biomarkers). | 3 years
  Variant S1P/S1PR related biomarkers; CIPN Questionnaire for Blood Collection Protocol (non-standardized questionnaire, 0-4 rating scales, 0 = no symptoms, 4 = very severe symptoms, symptoms: neuropathic pain severity/unpleasantness, sharpness, depth, tingling, numbness)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Lionberger, MD, PhD, Principal Investigator — St. Louis University